CLINICAL TRIAL: NCT03933124
Title: The Effect of Virtual Reality on Post-surgical Pain and Recovery.
Acronym: VIRTUAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL69077.091.19
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2020-10

CONDITIONS: Pain; Post-surgical Pain; Pain Management
Keywords: Post-surgical pain; Virtual Reality; Distraction
MeSH Terms: conditions — Pain; Pain, Postoperative; Agnosia

STUDY DESIGN:
Intervention Model Description: An explorative study using a randomized controlled parallel design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Intervention group (Experimental): The intervention group includes 60 patients who will use Virtual Reality for postoperative pain. Participants will use Virtual Reality minimal 10 minutes, minimal 3 times a day on the second, third and fourth day after surgery, on the general ward.
  * 20 participants will receive an Oculus Go immersive 3D nature videos, games, meditation videos, google earth experiences and sports games.
  * 20 participants will receive a Relaxmaker with 2D nature videos
  * 20 participants will receive CareVRx with 3D nature videos and meditation videos.
  Interventions: Device: Virtual Reality
- Control group (No Intervention): The control group receives standard postoperative care.

INTERVENTIONS:
Device: Virtual Reality — The Virtual Reality intervention is used for 10 minutes minimal 3 times a day on postoperative day 2-4.
  Other Names: Relaxmaker; Oculus Go; CareVRx
  Arms: Virtual Reality Intervention group

SUMMARY:
This study evaluates the effect of Virtual Reality (VR) on pain and recovery in 100 post-operative patients. 60 patients will be included in the intervention group; they will use VR minimal 3 times a day on day 2-4 after surgery, on the surgical ward, as an add-on intervention next to standard care. 40 patients in the control group will only receive standard postoperative care.

DETAILED DESCRIPTION:
Adequate management of post-surgical pain (PSP) may contribute to improved clinical and socioeconomic outcomes. Facilitating an adequate level of PSP relief is a challenging problem: the analgesics that are most frequently used, for example, opioids and non-steroidal anti-inflammatory drugs (NSAIDs), often come with side effects and do not always provide sufficient pain relief. Therefore, pain management is increasingly focusing on (additional) non-pharmacological analgesics, including Virtual Reality (VR).

VR immerses the user in a virtual world through a head mounted device (HMD). VR is, among other things, taught to be effective through distraction: it diverts attention away from the nociceptive input, resulting in less available attention for pain perception. In both clinical and experimental studies, VR has shown to be effective in reducing pain, anxiety and stress.

Although this distraction method is increasingly studied in the past years, VR pain relief has mostly been investigated as an intervention during painful procedures in specific research populations. For example, VR has been studied during wound dressing changes in burn wound patients in children and adolescents, during venipuncture in children or during dental treatments. Furthermore, most VR studies used VR as a single intervention, measuring pre-post differences in pain scores or used a cross over design with one VR session and one control session. It is interesting to know whether VR is effective in reducing postoperative pain during more than one VR session. More research is needed in larger trials evaluating a broad sample of the general population including elderly, as the common hospitalized patient is of an older age nowadays. Finally, it is important to evaluate the feasibility and acceptability of VR in postoperative patients and to know whether there are predictive factors to select patients who can mostly benefit from VR interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patient underwent surgery
* Patient reports a postoperative pain score ≥4 on the first postoperative day at the surgical ward and pain score should also be marked with 'pain is not acceptable'.
* At the day of recruitment, the estimated length of stay is at least 4 days after inclusion.
* Patient is willing and able to comply with the trial protocol.
* Patient is at least 16 years old on the day the informed consent form will be signed.

Exclusion Criteria:

* Patient suffers from delirium or acute confusional state.
* Patient has (a history of) dementia, seizure or epilepsy.
* Patient with severe hearing/visual impairment not corrected.
* Patient is placed in isolation.
* The skin of the patient's head or face is not intact (for example head wounds, psoriasis, eczema).
* Unplanned (re)admission to the intensive care unit (ICU).
* Inclusion in another trial to evaluate new ways of treating pain

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Mean Daily pain score (VAS, visual analogue scale) | day 1-4, the first four postoperative days on the surgical ward
  Pain on average in the last 24h. VAS (visual analogue scale): 0-100 mm, 0 is defined as "no pain at all", 100 is "the worst pain the patient can imagine".

SECONDARY OUTCOMES:
Time to 30% pain reduction compared to pain scores on postoperative day 1. | day 1-4, the first four postoperative days on the surgical ward.
  Time to 30% pain reduction compared to pain scores on postoperative day 1.
Mean Daily worst pain score (VAS) | day 1-4, the first four postoperative days on the surgical ward.
  Worst pain in the last 24h.
Effect of pain on mobility (NRS, Numeric Rating Scale) | day 1-4, the first four postoperative days on the surgical ward.
  NRS score (Numeric Rating Scale): 0-10. 0 is defined as "no pain at all", 10 is "the worst pain the patient can imagine".
Difference in pain scores pre- and post- VR intervention (VAS) | Day 2-4 on the surgical ward.
  Pain pre- and postintervention in the VR intervention group.
Quality of recovery -15 questionnaire. | day 1-4, the first four postoperative days on the surgical ward.
  Quality of recovery -15 questionnaire.
Mean Daily Anxiety score (VAS). | day 1-4, the first four postoperative days on the surgical ward.
  Anxiety on average in the last 24h.
Mean Daily Stress score (VAS) | day 1-4, the first four postoperative days on the surgical ward.
  Stress on average in the last 24h.
State-Trait Anxiety Inventory (STAI)-6 questionnaire. | day 1-4, the first four postoperative days on the surgical ward.
  State-Trait Anxiety Inventory (STAI)-6 questionnaire.
Difference in anxiety scores pre- and post- VR intervention. (VAS) | Day 2-4 on the surgical ward.
  Anxiety pre- and postintervention in the VR intervention group.
Difference in stress scores pre- and post- VR intervention. (VAS) | Day 2-4 on the surgical ward.
  Stress pre- and postintervention in the VR intervention group.
Difference in depression scores pre- and post- VR intervention. (VAS) | Day 2-4 on the surgical ward.
  Depression pre- and postintervention in the VR intervention group.
Analgesic use | day 1-4, the first four postoperative days on the surgical ward.
  Analgesic use (paracetamol, NSAIDs, opioids, use of add-on/escape medication, daily defined dose of opioid, days to removal of epidural analgesia or PCA (patient-controlled intravenous analgesia, morphine IV), days to converting from opioids to NSAIDs or paracetamol without opioids).
Feasibility of VR | Day 1-4 postoperative
  Questionnaire, interview
Patients acceptability | Day 1-4 postoperative
  Questionnaire, interview
Tolerability of Virtual Reality | Day 1-4 postoperative
  Questionnaire, interview

CONTACTS AND LOCATIONS:
Overall Officials: Harry van Goor, MD,PhD,FRCS, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical center, Nijmegen, Netherlands